CLINICAL TRIAL: NCT06776523
Title: Boosting Refugee Integration Through Psychological Intervention
Acronym: BRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-2023-00857
Record Dates: First submitted 2024-12-18; First posted 2025-01-15 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Psychological Distress; PTSD; Trauma; Common Mental Health Problems
Keywords: Problem Management Plus; Psychological Distress; Mental Health Care; Refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The RCT will inform us about the effectiveness of PM+ under usual practice conditions.
  After the screening and baseline assessment, thousand five hundred participants (N = 1500) will be involved in the RCT (assigned to either receiving the PM+ intervention right after the baseline assessment (N = 750) or twelve months later (N = 750)). Participants who scored below the K10 cut-off will be assigned to an observational control group receiving no intervention (N = 500).
Who Masked: Outcomes Assessor
Masking Description: All instruments and questions of the screening and baseline assessment will be assessed as an assisted self-assessment in the presence of a trained assessor fluent in the participant's mother tongue and blind to the allocation status of the participants.The follow-up assessments are administered either as an online self-assessment, as an assisted online self-assessment or as an self-assessment in presence. In either case, the trained assessors are blind to the allocation status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group (Experimental): The participants who are assigned to the intervention group will receive five sessions of PM+, a psychological intervention which has been developed by the WHO. PM+ is a short, transdiagnostic (i.e., not specifically aimed at treating a certain mental disorder) program aiming to reduce common mental health symptoms and improve psychosocial functioning. In addition, participants will receive three telephone booster sessions and are provided with handouts and homework reminders.
  Interventions: Behavioral: Problem Management Plus
- waitlist control group (Other): The control group will receive the augmented PM+ intervention 12 months after the baseline assessment.
  Interventions: Behavioral: Problem Management Plus
- observational control group (No Intervention): Participants who scored below 20 on the K10 will will only be part of the baseline assessments and receive no intervention.

INTERVENTIONS:
Behavioral: Problem Management Plus — Problem Management Plus (PM+) is a brief, psychological intervention program based on CBT techniques that are empirically supported and formally recommended by the WHO. The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, facing fears, and accessing social support. These elements have been recommended in recent WHO guidelines.
  Additionally, the original five PM+ sessions will be augmented in two ways. First, the participants will receive three 30-45-minutes telephone booster sessions 10, 22, and 34 weeks after the final original PM+ session. The second augmentation strategy involves handouts and homework reminders.
  Arms: Intervention group; waitlist control group

SUMMARY:
Refugees and asylum seekers (RAS) face numerous stressors and adversities which put them at risk for developing mental health problems. However, access to adequate mental health care in host countries is limited. To address this problem, the World Health Organization (WHO) introduced Problem Management Plus (PM+), a short, low-intensity psychological intervention administered by non-professionals, aiming to alleviate common mental disorders among crisis-affected communities.

The present study aims at expanding the existing PM+ intervention by providing additional booster sessions and homework reminders while evaluating its effectiveness and implementation in the public health system.

DETAILED DESCRIPTION:
Refugees and asylum seekers (RAS) are often exposed not only to potentially traumatic events before and during migration but also to significant post-migration stressors. Due to this combined burden, RAS are at increased risk for developing mental health problems. In accessing mental health care in the host countries, however, they face several barriers including waitlists, stigma and communication difficulties. Consequently, RAS are frequently underdiagnosed and often do not receive adequate medical treatment despite an urgent need.

To improve the access to evidence-based psychological interventions, the WHO developed a series of scalable interventions. One of these is Problem Management Plus (PM+), a brief, low-intensity psychological intervention, delivered by paraprofessionals, that addresses common mental disorders in people affected by adversity. PM+ consists of 5 sessions that comprise evidence-based techniques of (a) problem solving, (b) stress management, (c) behavioral activation, and (d) accessing social support. The present study aims at expanding the existing PM+ intervention by providing additional booster sessions and homework reminders.

PM+ has been proven to be an effective method for reducing mental health problems and improving the psychosocial functioning of people in crisis in various countries and contexts, including Switzerland.

Despite its effectiveness, far too little attention has been paid to the successful implementation of such low-intensity psychological interventions into real-world health care systems.

To address this gap, the present study aims to evaluate the effectiveness of augmented PM+ on mental health outcomes over 3 months under usual practice conditions and its implementation in the public health care system by using a pragmatic randomized clinical trial design.

ELIGIBILITY:
The inclusion criteria for participating in the study are:

* refugees and asylum seekers (RAS) aged 16 or older;
* residing in one of the participating local sites (Swiss municipalities, namely, Gemeinden, and transitional asylum centers, namely, Durchgangszentren) where PM+ is offered and which gave their consent for participation in the RCT;
* speaking at least one of the following 12 languages: German, English, French, Arabic, Farsi, Kurdish, Tigrinya, Turkish, Ukrainian, Russian, Tamil, and Pashto;
* obtaining a score of 20 or higher on the Kessler Psychological Distress Scale (K10; Kessler et al., 2002), a brief clinically validated screening questionnaire that assesses general psychological distress in the past 30 days. A score equal to or higher than 20 is used as an indication of moderate to high levels of psychological distress.

The exclusion criteria for participating in the study are:

* significant cognitive or neurological impairment measured through specific tools developed by the WHO and integrated into the PM+ manual (impairment questionnaire);
* acute medical conditions or severe mental disorders (e.g., psychotic or substance-abuse disorders) measured through specific tools developed by the WHO and integrated into the PM+ manual (impairment questionnaire);
* acute risk of suicide as measured by the Suicidal Ideation Attribution Scale (SIDAS; van Spijker et al., 2014) and the Thoughts of Suicide Questionnaire (World Health Organization WHO, 2016).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in psychological distress | Baseline assessment, 3 month FU assessment (3 months after baseline)
  Change in psychological distress will be measured with the Hopkins Symptom Checklist (HSCL-25). Items are rated on a scale from 1 to 4. Higher scores indicate more pronounced symptom severity.

SECONDARY OUTCOMES:
Change in psychological distress | 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after baseline), 24 month FU assessment (24 months after b.), 36 months FU (36 months after b.)
  Change in psychological distress will be measured with the Hopkins Symptom Checklist (HSCL-25). Items are rated on a scale from 1 to 4. Higher scores indicate more pronounced symptom severity.
Change in posttraumatic stress disorder symptoms | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after b.), 24 month FU assessment (24 months after b.), 36 months FU (36 months after b.)
  Change in posttraumatic stress disorder symptoms will be assessed using the 4-item short form of the PCL-5. Items are rated on a scale from 0 to 4 with higher scores indicating more pronounced symptom severity.
General psychological distress | Screening, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after baseline)
  General psychological distress will be measured with the Kessler Psychological Distress Scale (K10), a brief screening questionnaire assessing general psychological distress in the past 30 days. It consists of ten items (e.g., "During the last 30 days, about how often did you feel tired out for no good reason?") rated on a 5-point Likert scale (1 = "none of the time" to 5 = "all of the time"), before summation (range 10-50).
Somatic symptoms | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after b.), 24 month FU assessment (24 months after b.), 36 months FU (36 months after b.)
  Somatic symptoms will be assessed using the Somatic Symptom Scale (SSS-8). Items are rated on a scale from 0 to 4 with higher scores indicating higher symptom severity.
Reduction of post-migration stressors | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after b.), 24 month FU assessment (24 months after b.), 36 months FU (36 months after b.)
  Changes in post-migration stressors will be assessed using a 9-item version of the Post Migration Living Difficulties Checklist (PMLDC). Items are rated on a scale from 0 to 4 with lower scores representing fewer post-migration stressors.
Exposure to potentially traumatic events | Baseline assessment
  Exposure to potentially traumatic events is indexed using a list of seven traumatic experiences. Overall trauma exposure is represented by a count of the number of traumatic event types (ranging from 0 to 7) experienced by each participant; higher scores indicate experience of more forms of traumatic events.
Level of integration | Baseline assessment, 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after b.), 24 month FU assessment (24 months after b.), 36 months FU (36 months after b.)
  Level of integration will be measured using the Immigration Policy Lab Integration Index (IPL-24).
Suicidal Ideation | Screening, 6 month follow-up assessment (6 months after baseline), 36 month follow-up assessment (36 months after baseline)
  Suicidal Ideation is measured using the Suicidal Ideation Attribution Scale (SIDAS), a brief measure of severity of suicidal ideation assessing frequency, controllability, closeness to attempt, level of distress associated with the thoughts and impact on daily functioning. It consists of five items rated on a 11-point scale (0 = "Never" to 10 = "Always").
Self-efficacy | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after baseline)
  Self-efficacy is assessed using a subscale of the Compound Psychological Capital Scale (CPS). This subscale consists of three items (e.g., "I can solve most problems if I invest the necessary effort") of the General Self-Efficacy Scale (GSE). Each item is rated on a 6-point Likert type scale ranging from 1 = "strongly disagree" to 6 = "strongly agree".
Prolonged Grief | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after baseline)
  Prolonged Grief will be assessed using a slightly adapted version of the Prolonged Grief Disorder Scale (PG-13). The items are rated on a scale from 1 to 5 with higher scores more pronounced symptom severity.
Assessing the extent to which the strategies taught in PM+ are used before and after the study participation with the Reducing Tension Checklist | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after baseline)
  The outcome is measured with a nine-item scale that was developed to assess the extent to which the participants perceives that they use the specific strategies, which are trained during the study intervention. The items are rated on a scale from 0 to 4. Higher scores represent greater usage of the strategies.
Anger | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment (12 months after baseline), 24 month FU assessment (24 months after b.), 36 months FU (36 months after b.)]
  Anger will be assessed using the Dimensions of Anger Reactions Questionnaire (DAR-5). The 5 items are rated on scale from 1 to 5 with higher scores indicating worse symptomatology.
Time and risk preferences | Baseline assessment, 3 month FU assessment (3 months after baseline)
  Time and risk preferences are assessed using five questions of the Global Preference Survey (GPS), an experimentally validated survey measure. It consists of one self-assessment question (rated on a scale from 0 to 10 with higher scores indicating a greater preference) and a 4-item series of interdependent binary choices between immediate and delayed financial rewards, a format commonly referred to as a "staircase" procedure. In each of the binary choice question, participants must decide between receiving a payment today or a larger payment in twelve months (time preference) or between a sure choice and a lottery (risk preference).
Facial Expression | Baseline assessment, 3 month FU assessment (3 months after baseline)
  After responding to questions about positive / negative past and imagined future experiences, participants are asked to rate the emotionality of the experience they had during the speech on a 10-point scale (1 = not at all distressing, 10 = extremely distressing). Analyses will be conducted to calculate facial actions, acoustic quality, and speech content using the OpenDBM software.
Assessment of Coping Strategies | Baseline assessment, 3 month FU assessment (3 months after baseline)
  Participants will also be asked about current life stressors and how they cope with these stressors. Analyses will be conducted to calculate facial actions, acoustic quality, and speech content using the OpenDBM software.
Counterfactual Comparisons | Baseline assessment, 3 month FU assessment (3 months after baseline)
  To assess counterfactual comparisons regarding well-being, two items of the Comparison Standards Scale for Well-being (CSS-W) will be used. The two items of the CSS-W ask about frequency of well-being comparisons in the past three weeks on six-point Likert scales (0 = not at all to 5 = very often).

OTHER OUTCOMES:
Use of health care services and medications | Two years before (or since arrival in Switzerland if less than two years) to four years after study inclusion
  Investigators will complement the self-reported survey-based health measures with register data from the major health insurance providers in Switzerland covering the RAS population to explore the use and involved costs of health care services and medications.
Impact of asylum process on mental health | Two years before (or since arrival in Switzerland if less than two years) to four years after study inclusion
  To explore the consequences of the length of the asylum process on mental health outcomes (and the potential of PM+ to alleviate them), register information on the length of the asylum process, defined as the days between the submission of the asylum application and the date of the (initial) decision by the State Secretariat of Migration (SEM), will be used.
Labour market integration | Two years before (or since arrival in Switzerland if less than two years) to four years after study inclusion
  To assess labour market integration investigators will leverage data from the AHV-insurance to obtain information on participants' employment, considered a sign of successful integration in the labour market. The data indicates periods of employment and levels of earnings for each individual working in Switzerland.
Impact of residence status | Two years before (or since arrival in Switzerland if less than two years) to four years after study inclusion
  To assess the impact of residence status, population and household data will be obtained which records movements within Switzerland, individuals' resident status and changes of the latter. They are important factors impacting mental health and integration that need to be included in the analysis.
Impact of cantonal regulations | Two years before (or since arrival in Switzerland if less than two years) to four years after study inclusion
  The impact of cantonal regulations will be assessed using register data which provides up to date information on cantonal variation regulating labour market access, including length of the initial employment bans, occupational and mobility restrictions.
Integration | Two years before (or since arrival in Switzerland if less than two years) to four years after study inclusion
  To assess integration of RAS population, population and household data will be used. This database provides indicators of integration, including marriages between foreign and Swiss residents, and naturalization, which complements the study's integration outcomes with more accurate measures, as compared to the self-reported data.

CONTACTS AND LOCATIONS:
Overall Officials: Naser Morina, PD Dr., Principal Investigator — Klinik für Konsiliarpsychiatrie und Psychosomatik
Locations (1):
- Klinik für Konsiliarpsychiatrie und Psychosomatik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaaij J, Kiselev N, Berger C, Bryant RA, Cuijpers P, de Graaff AM, Fuhr DC, Hemmo M, McDaid D, Moergeli H, Park AL, Pfaltz MC, Schick M, Schnyder U, Wenger A, Sijbrandij M, Morina N. Feasibility and acceptability of Problem Management Plus (PM+) among Syrian refugees and asylum seekers in Switzerland: a mixed-method pilot randomized controlled trial. Eur J Psychotraumatol. 2022 Jan 31;13(1):2002027. doi: 10.1080/20008198.2021.2002027. eCollection 2022. PMID 35126880
- [Background] de Graaff AM, Cuijpers P, Twisk JWR, Kieft B, Hunaidy S, Elsawy M, Gorgis N, Bouman TK, Lommen MJJ, Acarturk C, Bryant R, Burchert S, Dawson KS, Fuhr DC, Hansen P, Jordans M, Knaevelsrud C, McDaid D, Morina N, Moergeli H, Park AL, Roberts B, Ventevogel P, Wiedemann N, Woodward A, Sijbrandij M; STRENGTHS Consortium; STRENGTHS consortium. Peer-provided psychological intervention for Syrian refugees: results of a randomised controlled trial on the effectiveness of Problem Management Plus. BMJ Ment Health. 2023 Feb;26(1):e300637. doi: 10.1136/bmjment-2022-300637. Epub 2023 Feb 8. PMID 36789918
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Steel Z, Chey T, Silove D, Marnane C, Bryant RA, van Ommeren M. Association of torture and other potentially traumatic events with mental health outcomes among populations exposed to mass conflict and displacement: a systematic review and meta-analysis. JAMA. 2009 Aug 5;302(5):537-49. doi: 10.1001/jama.2009.1132. PMID 19654388